CLINICAL TRIAL: NCT06590623
Title: The Effect of Acute Exogenous Oral Ketone Supplementation on Immune Cells Function and Immune Cells Histone Β-hydroxybutyrylation
Acronym: Acute_Ketone
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Jonathan Little, Professor, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: H24-02548
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Ketosis, Metabolic; Immune Functions; Histone Deacetylase (HDAC) Activity
Keywords: Ketone supplement; Exogenous ketones; Immune function; β-hydroxybutyrylation; Beta-Hydroxybutyrate
MeSH Terms: conditions — Ketosis; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- exogenous ketone supplement (Experimental): Participants will consume a ketone monoester supplement (KetoneAid KE4) at a dose of 0.75 g/kg of body weight.
  Interventions: Dietary Supplement: Ketone Monoester (KE)

INTERVENTIONS:
Dietary Supplement: Ketone Monoester (KE) — Participants will receive an exogenous ketone supplement (KetoneAid KE4) in a fasted state in the morning, at a dosage of 0.75 g/kg of body weight.
  Other Names: Exogenous ketone

SUMMARY:
To conduct a single-arm pilot study to determine how acute ingestion of an exogenous ketone monoester supplement alters the histone lysine β-hydroxybutyrylation and immune function in healthy human monocytes and lymphocytes.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 19
* Able to fast overnight

Exclusion Criteria:

* Being a competitive endurance athlete.
* Following a ketogenic diet, low-calorie diet, periodic fasting regimen, or regularly consuming ketogenic supplements.
* Being unable to travel to and from the university
* Being pregnant.
* Having been diagnosed with a chronic disorder of glucose or fat metabolism, including type 2 diabetes, chronic pancreatitis, or gallbladder disease
* Being unable to read or communicate in English.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
β-hydroxybutyrylation of histone in human immune cells using Western blotting | Before (fasted state) and 2 hours after the consumption of the exogenous ketone supplement.
  The β-hydroxybutyrylation of histones in human monocytes and lymphocytes will be assessed before and 2 hours after the consumption of an exogenous ketone supplement. Protein samples will be collected from the cells, and the levels of histone β-hydroxybutyrylation will be quantified using Western blotting.

SECONDARY OUTCOMES:
Change in beta-hydroxybutyrate concentration | Capillary beta-hydroxybutyrate will be measured before, 30, 60, 90, 120 and 180 minutes after the consumption of exogenous ketone supplement.
  Capillary beta-hydroxybutyrate concentration will be measured using FreeStyle Neo β ketone test before, 30, 60, 90, 120, and 180 minutes after the consumption of exogenous ketone supplement.
Change in glucose concentration | Capillary glucose concentration will be measured before, 30, 60, 90, 120, and 180 minutes after the consumption of exogenous ketone supplement.
  Capillary glucose concentration will be measured using FreeStyle Neo glucose test before, 30, 60, 90, 120, and 180 minutes after the consumption of exogenous ketone supplement.
Change in blood pressure | Before, 30, 60, 90, 120 and 180 minutes after the consumption of the exogenous ketone supplement.
  Systolic and diastolic blood pressure will be measured using an automatic blood pressure device before, and at 30, 60, 90, 120, and 180 minutes after consuming the exogenous ketone supplement.
Change in resting heart rate | Before, 30, 60, 90, 120 and 180 minutes after the consumption of the exogenous ketone supplement.
  Resting heart rate will be measured using continuous heart rate measurement (POLAR H10) before, and at 30, 60, 90, 120, and 180 minutes after consuming the exogenous ketone supplement.
Alteration in immune cell functions | Before (fasted state) and 2 hours after the consumption of the exogenous ketone supplement.
  Immune cell functions in healthy individuals will be assessed using whole blood and monocyte cultures treated with lipopolysaccharide (with or without interleukin-10) and the subsequent measurement of cytokine secretion (e.g., TNF-a), both before and 2 hours after the ingestion of a ketone supplement.
Monocytes and lymphocytes Immunophenotyping | Before (fasted state) and 2 hours after the consumption of the exogenous ketone supplement.
  Immunophenotyping of monocytes and lymphocytes will be conducted by assessing surface receptor expression using flow cytometry. Various antibodies will be used, including CD14, CD16, and TLR4 for monocytes, and CD4 and CD8 for lymphocytes, at baseline and 2 hours following the ingestion of a ketone supplement.
Gastrointestinal Disturbance | Before, and at 30, 60, 90, 120, and 180 minutes after consuming the exogenous ketone supplement.
  Gastrointestinal disturbance will be measured using a 10-cm visual analogue scale to assess nausea, urge to vomit, bloating, belching, and cramps before, and at 30, 60, 90, 120, and 180 minutes after consuming the exogenous ketone supplement. A higher score, closer to the right end of the 10-cm visual analogue scale, indicates greater gastrointestinal disturbance.

CONTACTS AND LOCATIONS:
Locations (1):
- University of British Columbia Okanagan Campus, Kelowna, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared to ensure the privacy and confidentiality of participants, in accordance with ethical guidelines and data protection regulations. Additionally, this was not included in the informed consent, which did not cover data sharing or address potential risks of re-identification.